CLINICAL TRIAL: NCT00354809
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Effects of Morning Administration of GW679769 (10mg and 30 mg) on Polysomnograph Sleep Recordings, Subjective Sleep Assessment, Daytime Cognition and Psychomotor Function in Subjects With Primary Insomnia
Brief Title: Evaluation of A Morning Dosing Of A New Medicine And Its Effects On Sleep At Bedtime In Subjects With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MAD105516
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Sleep Initiation and Maintenance Disorders; Insomnia
Keywords: cognition; Primary Insomnia; sleep; polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769

SUMMARY:
This study is designed to determine whether morning doses of GW679769, taken daily for 1 to 9 days, will promote sleep during the following night without significant post-dose thinking impairment and drowsiness in subjects with primary insomnia.

ELIGIBILITY:
Inclusion criteria:

* Difficulty going to sleep and/or staying asleep during at least the past 3 months.
* Insomnia must result in significant distress or impairment in functioning at home, socially or at work.
* Otherwise good health with no significant or unstable medical disorder including psychiatric, neurological, endocrine, heart, lung or gastrointestinal disorders, drug/alcohol abuse, cognitive impairment, cancer or chronic pain conditions such as arthritis.

Exclusion criteria:

* History of other sleep disorders such as sleep apnea or restless leg syndrome; regular sleep habits, including bedtime between 9 PM and midnight, nightshift/rotating shift work, frequent napping or planned travel across >2 time zones.
* Use to moderate use of nicotine, caffeine and alcoholic products.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Comparison of GW679769 and placebo when taken daily in the morning, on the time needed to fall asleep at bedtime on Days 1/2 and 8/9 of treatment, as assessed at a sleep clinic. | 9 Days

SECONDARY OUTCOMES:
Comparison of GW679769 and placebo on total sleep time and time awake after initial sleep onset on Days 1/2 and 8/9 of treatment, as assessed at a sleep clinic. Daily sleep questionnaires and mental functioning tests on Days 1 and 9 of treatment. | 9 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (13):
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Hinesville, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
- France (3):
  - GSK Investigational Site, Clamart
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouffach
- Germany (5):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Schwalmstadt, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Berlin, State of Berlin